CLINICAL TRIAL: NCT04470388
Title: A Phase 1b Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of EDP 514 in Viremic Chronic Hepatitis B Virus Infected Patients Not Currently on Treatment
Brief Title: A Study of EDP-514 in Patients With Chronic Hepatitis B Virus Infection Who Are Not Currently on Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP 514-002
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Chronic HBV Infection
Keywords: Multiple Ascending Dose; hepatitis B virus; HBV
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDP-514 HBV MAD Cohorts (Experimental): EDP-514 capsule Dose 1, Dose 2 and Dose 3 orally, once daily for 28 days.
  Interventions: Drug: EDP-514
- EDP-514 HBV MAD Placebo Cohort (Placebo Comparator): Matching placebo, orally, once daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-514 — Oral Capsule
  Arms: EDP-514 HBV MAD Cohorts
Drug: Placebo — Placebo to match EDP-514
  Arms: EDP-514 HBV MAD Placebo Cohort

SUMMARY:
This is a randomized, double-blind, placebo-controlled study in viremic chronic hepatitis B subjects, assessing the safety, tolerability, pharmacokinetics and antiviral activity of 28 Days treatment with EDP-514.

DETAILED DESCRIPTION:
The study assesses multiple ascending doses of EDP-514 compared to placebo for 28 days in viremic chronic CHB-infected subjects not currently on treatment.

Each cohort will enroll a total of 8 subjects who will be randomized to receive EDP-514 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 70 years, inclusive
* HBV DNA levels:

  * For subjects who are HBeAg positive at Screening, a Screening HBV DNA level in serum/plasma that is ≥20,000 IU/ml, or
  * For subjects who are HBeAg negative at Screening, a Screening HBV DNA level in serum/plasma that is ≥2,000 IU/mL, and
  * For all subjects, no HBV DNA serum/plasma test values <1,000 IU/ml over the previous 12 months (using an approved test)
* CHB subjects must not have been on prescribed anti-HBV treatment for at least 12 months prior to Screening

Exclusion Criteria:

* A documented prior diagnosis of cirrhosis
* Pregnant or nursing females
* Coinfection with human immunodeficiency virus (HIV), HCV, HDV, HAV, or HEV
* Chronic liver disease of a non-HBV etiology; coexisting liver or biliary diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events | Up to 84 Days in HBV MAD Cohorts

SECONDARY OUTCOMES:
Cmax of EDP-514 | Up to 28 Days in HBV MAD Cohorts
AUC of EDP-514 | Up to 28 Days in HBV MAD Cohorts
Change from baseline in HBV DNA Viral Load Assay | through Day 28 in HBV MAD Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (10):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Taiwan (9):
  - Chia-Yi Christian Hospital, Chiayi City, Chiayi
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital/E-DA Cancer Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation, Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District